CLINICAL TRIAL: NCT04476433
Title: Application of a Program in Chronic Pediatric Patients With Different Pathologies and in Their Families.
Brief Title: Intervention in Chronic Pediatric Patients and Their Families.
Acronym: FACTORADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital General Universitario de Valencia (Other); Hospital Clínico Universitario de Valencia (Other); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FACTORADAPT
Record Dates: First submitted 2020-07-03; First posted 2020-07-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes; Allergic Rhinitis; Allergic Asthma; Asthma; Short Stature; Food Allergy; Atopic Dermatitis; Rhinoconjunctivitis; Cystic Fibrosis; Primary Ciliary Dyskinesia; Pulmonary Disease
Keywords: Caregivers; Adolescent; Anxiety; Depression; Quality of life; Intervention Study
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Rhinitis, Allergic; Asthma; Dwarfism; Food Hypersensitivity; Dermatitis, Atopic; Cystic Fibrosis; Ciliary Motility Disorders; Lung Diseases; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients and caregivers who receive the treatment program, will previously constitute their own control group (waiting list control group).
- Experimental Group (Experimental): Patients and caregivers who receive the treatment program, will previously constitute their own control group (waiting list control group). Thus, diagnostic measures will be obtained in all of them in an initial evaluation (T1), and after 6 months of this evaluation the treatment program will be started. In the first contact session at 6 months after T1 all subjects (patients and relatives) will be re-evaluated (T2) and after this the treatment program will be started (within an estimated time of 15 days maximum from this second pre-treatment evaluation, the estimated duration of treatment being 5 months). After the completion of the patient and family treatment sessions, a new diagnostic test pass will be performed (T3) (within an estimated maximum period of 15 days from the completion of treatment) in order to evaluate the post-treatment change. Thus, the estimated time between T2 and T3 will be equivalent to that between T1 and T2, being 6 months.
  Interventions: Other: Ten Vida (10Vida)

INTERVENTIONS:
Other: Ten Vida (10Vida) — 10Vida is a psychoeducational and emotional programme for chronic illness in adolescents and their families.
  Arms: Experimental Group

SUMMARY:
This project consists of a psychological intervention in patients and their families with different chronic diseases in order to carry out a comparative study between medical pathologies to know which are the protective or risk variables for the adaptation to the disease.

DETAILED DESCRIPTION:
Adolescence is a period characterized by a multitude of changes at the biopsychosocial level, all of which also implies many challenges. If the diagnosis or the presence of a chronic disease or condition (CD) is added, the adjustment of the adolescent to this period become even more difficult.

The World Health Organization (WHO) (2017) defines chronic diseases (CD) as "long-lasting and usually slow-progressing diseases". Among the main child-juvenile CDs are the allergic, the endocrine; in particular, Diabetes Mellitus Type 1 (DM1) and Short stature (SS), and respiratory, such as bronchial asthma (BA).

Chronic pediatric disease is a medical condition that affects both the patient and the family caregiver. Chronic disease is characterized by unforeseeable changes in the course of the disease, a reduction in physical capacity, changes in appearance, a prolonged dependence on medical specialists, continuous treatments and the need for assistance.

The presence of CD in adolescence is a risk factor for developing a psychological disorder. The most common psychopathology in childhood-juvenile CD is emotional, particularly anxiety symptoms, followed by depression symptoms, being possible the development of an anxiety disorder or of a major depression.

When someone is diagnosed with a chronic disease, the family as a whole is affected by the stressors associated with the disease and the side effects of treatment, being inevitable the alteration of the whole family system, especially in cases where the patient is a infant or adolescent. In addition, it is necessary to underline that studies indicate that most of the care of adolescent patients generally is undertaken by one specific member of the family, usually called the main caregiver. The stress due to the care tasks has been associated with anxiety and depression symptoms, often causing emotional disturbances in the caregivers, associating the above with greater emotional symptomatology in adolescents and worse control of their disease.

That's why more studies like the one proposed are needed to study more deeply the protective factors of psychological and physical health during the course of chronic disease at this stage of life, both in the adolescent patients as well as in their family.

The main aim of this research is to study the psychosocial factors, adjustment to the disease and improvement of psychological well-being in the adolescent population with chronic disease. In order to do this, the investigators are going to analyse the main characteristics (psychological, family related and adjustment to disease) in the adolescent population with endocrinological problems (short stature and diabetes mellitus type 1), respiratory (asthma) and allergenic problems. These characteristics will also be analysed in the family of the adolescent patients. The personal adaptation profiles and families features that favor the psychological and physical health in these patients and their family caregivers will be also identified. In addition, the investigators also propose as an aim the development and implementation of an assessment and intervention program (in a pilot sample) that provides socio-emotional education in adolescent patients with chronic disease and their family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis at least 6 months.
* To have signed the informed consent.

Exclusion Criteria:

* No previous psychological diagnosis.
* Attention Deficit Hyperactivity Disorder(ADHD), epilepsy or brain tumor
* Infant cerebral palsy
* Not understanding the Spanish language

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change Emotional Distress in caregivers (Baseline-Pre-Post) | Baseline up to 12 months
  Assessment with Hospital Anxiety and Depression Scale in caregivers (HADS): Screening instrument for the detection of affective disorders, in non-psychiatric subjects who go to hospitals. The scale is made up of 14 items, with a range of scores from 0 to 42. The interpretation is that the higher the score, the greater the presence of anxiety-depressive symptoms.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change Emotional Distress in patients (Baseline-Pre-Post) | Baseline up to 12 months
  Assessment with Hospital Anxiety and Depression Scale in patients (HADS): Screening instrument for the detection of affective disorders, in non-psychiatric subjects who go to hospitals. The adaptation for this sample, it is made up of 11 items, with a range of scores from 0 to 33. The interpretation is that the higher the score, the greater the presence of anxiety-depressive symptoms.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change Caregiver burden (Baseline-Pre-Post) | Baseline up to 12 months
  Assessment with Parental Inventory: It aims to assess the stress of parents with children who require regular medical attention. It consists of 12 situations related to the hospital environment that are considered potentially stressful for parents with sick children. The range of scores is 12 to 60. And it is interpreted like higher scores, higher levels of stress.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change Emotional competences in patients (Baseline-Pre-post) | Baseline up to 12 months
  Emotional Skills and Competence Questionnaire (ESCQ-21): this is a self-report measure developed by Takšić to assess emotional competence. In the present study, the reduced version (ESCQ-21) was used, adapted and validated in a Spanish sample by Schoeps et al. The aim of assessing is emotional competence: perception and comprehension, expressing and labeling and management and regulation)
Change Self-esteem in patients (Baseline-Pre-Post) | Baseline up to 12 months
  Rosenberg Self-Esteem Questionnaire. It assesses the level of self-esteem. It is made up
Change of Perceived level of disease threat (Baseline-Pre-Post) | Baseline up to 12 months
  Brief Disease Perception Questionnaire (B-IPQ): This is a measure of patients' cognitive

SECONDARY OUTCOMES:
Change Resilience in caregivers (Baseline-Pre-Post) | Baseline up to 12 months
  Connor-Davidson Resilience Scale to assess the ability to cope with stress and adversity. The resilience scale is made up of 10 items, with a range of scores from 0 to 40, with higher scores indicating greater resilience.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change of Adaptation to chronic disease (DM1) (Baseline-Pre-Post) | Baseline up to 12 months
  Adaptive response questionnaire to the disease in diabetic patients: with the aim of evaluating the elements involved in the psychological and social response in pediatric diabetic patients. This instrument includes cognitive, emotional and behavioural elements that may be related to the adjustment response to the disease. The lower the score, the more severe the disease, the worse the health behaviour, the various complaints associated with the disease.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change of Adaptation to chronic disease (Respiratory chronic diseases) (Baseline-Pre-Post | Baseline up to 12 months
  This questionnaire evaluates health-related quality of life in relation to chronic respiratory problems. It is made up of 4 dimensions: sensation of dyspnea, sensation of fatigue, emotional symptomatology and disease control.
  The total score is obtained by adding up the score in each of the dimensions and dividing by 4. The resulting evaluation ranges from 1 (maximum affectation of up to 7 (no affectation) First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change of Adaptation to chronic disease (Rhinoconjunctivitis) (Baseline-Pre-Post) | Baseline up to 12 months
  It is a specific quality of life assessment instrument for the pediatric population with rhinoconjunctivitis. It aims to obtain a measure of the impact that allergic symptoms have on patients' daily functioning, and not only the severity and frequency. All items are weighted equally and a higher score is indicative of a poorer quality of life.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change of Adaptation to chronic disease (Food Allergy)(Baseline-Pre-Post) | Baseline up to 12 months
  Quality of Life Questionnaire in Food Allergy (FAQLQ- TF) It assessed quality of life relation with food allergy. The range of scores is from 0 to 6. The interpretation of the scores is reversed, i.e. the lower the score, the better the perceived quality of life.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 months after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 months after the second measurement the third measurement of the same variable was carried out.
Change in family functioning in caregivers (Baseline-Pre-Post) | Baseline up to 12 months
  Family Functioning Questionnaire (CAF) based on Olson's model. It was created with the aim of constructing a measuring instrument to evaluate the variables that make up the dynamics of a family
Change in parental styles in patients (Baseline-Pre-Post) | Baseline up to 12 months
  Scale for the evaluation of the educational style of parents of adolescents (EP). It allows evaluating the perception that adolescents have of the educational style of their parents.
Change Psychological well-being (Baseline-Pre-Post) | Baseline up to 12 months
  Psychological well-being scale for adolescents (BIEPS-J) to determine the level of psychological well-being in adolescents

OTHER OUTCOMES:
Glycaemic control (Baseline-Pre-Post) | Baseline up to 12 months
  HbA1c: It will be used to evaluate the glycemic control of the diabetic patient in endocrinology diseases
Weight (Baseline-Pre-Post) | Baseline up to 12 months
  Kilograms For assessment of nutritional status
Height (Baseline-Pre-Post) | Baseline up to 12 months
  Meters For assessment of nutritional status
Body mass index (BMI) (Baseline-Pre-Post) | Baseline up to 12 months
  BMI in kg/m^2, for assessment of nutritional status
Spirometry values (Baseline-Pre-Post) | Baseline up to 12 months
  All values obtained are expressed as volume (in ml). The main spirometric parameters recorded are forced vital capacity (FVC), vital capacity (VC), peak expired air volume in the first second (FEV1) and peak expiratory flow (PEF).
Blood test ( Baseline-Pre-Post) | Baseline up to 12 months
  For monitoring nutritional status (blood concentration of protein, lipids, fat-soluble vitamins, iron and calcium-phosphorus metabolism) and blood concentration of c) glucose metabolism d) acute phase reactants and immune status (immunoglobulins, alpha1 antitrypsin, and e) hepatic and renal functions.) exocrine pancreatic function
  • glucose metabolism d) acute phase reactants and immune status (immunoglobulins, alpha1 antitrypsine)
Exocrine pancreatic test ( Baseline-Pre-Post) | Baseline up to 12 months
  For monitoring pancreatic test, faecal elastase and steatorrhoea, and hepatic and renal functions.

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez-Marín, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No